CLINICAL TRIAL: NCT00143234
Title: Clinical Utility of Amlodipine/Atorvastatin to Improve Concomitant Cardiovascular Risk Factors of Hypertension and Dyslipidemia
Brief Title: Amlodipine/Atorvastatin Combination to Reduce the Health Risk of High Blood Pressure and High Cholesterol Levels
Acronym: GEMINI-AALA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Organization: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A3841024
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Hypertension; Hyperlipidemia
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Amlodipine

INTERVENTIONS:
Drug: Amlodipine/atorvastatin single pill

SUMMARY:
The purpose of the study is to measure the effect of the amlodipine/atorvastatin combination pill in reducing both elevated blood pressure and cholesterol levels to levels suggested by guidelines

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of both elevated blood pressure and low density lipoprotein cholesterol levels, requiring medication

Exclusion Criteria:

* Patients with blood pressure adequately maintained at goal with or without medication
* Patients currently treated with both amlodipine and atorvastatin or not at blood pressure or lipid level while taking the highest dose of amlodipine or atorvastatin, respectively

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1825
Dates: Start 2004-05; Study Completion 2005-07

PRIMARY OUTCOMES:
To evaluate the efficacy of amlodipine/atorvastatin therapy by assessing the percentage of intent-to-treat subjects achieving both BP and lipid treatment goals (JNC VII and NCEP ATP III)

SECONDARY OUTCOMES:
To assess changes from baseline in lipid profile and systolic and diastolic BP after 14 weeks treatment; and in this secondary and the primary objectives stratified by prior BP and lipid therapy, and in diabetic subjects; safety

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (96):
- Pfizer Investigational Site, Buenos Aires, Argentina
- Australia (7):
  - Pfizer Investigational Site, St Leonards, New South Wales
  - Pfizer Investigational Site, Southport, Queensland
  - Pfizer Investigational Site, Woolloongabba, Queensland
  - Pfizer Investigational Site, Heidelberg, Victoria
  - Pfizer Investigational Site, Melbourne, Victoria
  - Pfizer Investigational Site, Prahran, Victoria
  - Pfizer Investigational Site, Fremantle, Western Australia
- Brazil (7):
  - Pfizer Investigational Site, Belo Horizonte, Minas Gerais
  - Pfizer Investigational Site, Recife, Pernambuco
  - Pfizer Investigational Site, Botucatu, São Paulo
  - Pfizer Investigational Site, Campinas, São Paulo
  - Pfizer Investigational Site, Ribeirão Preto, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
  - Pfizer Investigational Site, SÃ£o Paulo, São Paulo
- Chile (2):
  - Pfizer Investigational Site, Santiago, RegiÃ³n Metropolitana
  - Pfizer Investigational Site, Santiago, RM
- Pfizer Investigational Site, Guatemala City, Guatemala
- Hong Kong (2):
  - Pfizer Investigational Site, Pokfulam Road
  - Pfizer Investigational Site, Sai Ying Pun
- India (6):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Mumbai, Nagpada Junction
  - Pfizer Investigational Site, New Delhi
- Indonesia (2):
  - Pfizer Investigational Site, Jakarta
  - Pfizer Investigational Site, Surabaya
- Israel (4):
  - Pfizer Investigational Site, Jerusalem
  - Pfizer Investigational Site, Rehovot
  - Pfizer Investigational Site, Tel Aviv
  - Pfizer Investigational Site, Tel Litwinsky
- Pfizer Investigational Site, Amman, Jordan
- Pfizer Investigational Site, Sasat, Kuwait
- Pfizer Investigational Site, Beirut, Lebanon
- Malaysia (4):
  - Pfizer Investigational Site, Kubang Kerian, Kelantan
  - Pfizer Investigational Site, Seremban, Negeri Sembilan
  - Pfizer Investigational Site, Kuching, Sarawak
  - Pfizer Investigational Site, Kuala Lumpur
- Mexico (6):
  - Pfizer Investigational Site, México, D.F
  - Pfizer Investigational Site, Aguascalientes
  - Pfizer Investigational Site, Metepec
  - Pfizer Investigational Site, México
  - Pfizer Investigational Site, Puebla City
  - Pfizer Investigational Site, San Luis Potosí City
- Pfizer Investigational Site, Casablanca, Morocco
- Pakistan (4):
  - Pfizer Investigational Site, Peshawar, Khyber Pakhtunkhwa
  - Pfizer Investigational Site, Faisalabad, Punjab Province
  - Pfizer Investigational Site, Islamabad, Punjab Province
  - Pfizer Investigational Site, Lahore, Punjab Province
- Pfizer Investigational Site, Lima, Peru
- Philippines (5):
  - Pfizer Investigational Site, San Juan City, National Capital Region
  - Pfizer Investigational Site, Phippine General Hospital, Taft Avenue, Manila City
  - Pfizer Investigational Site, Filinvest, Alabang
  - Pfizer Investigational Site, Manila
  - Pfizer Investigational Site, Quezon City
- Saudi Arabia (2):
  - Pfizer Investigational Site, Khobar
  - Pfizer Investigational Site, Riyadh
- Pfizer Investigational Site, Singapore, Singapore
- South Africa (8):
  - Pfizer Investigational Site, Worcester, Cape Province
  - Pfizer Investigational Site, Arcadia, Pretoria, Gauteng
  - Pfizer Investigational Site, Midrand, Johannesburg, Gauteng
  - Pfizer Investigational Site, Sunnyside, Pretoria, Gauteng
  - Pfizer Investigational Site, Chatsworth, KwaZulu-Natal
  - Pfizer Investigational Site, Kwa-Zulu Natal, KwaZulu-Natal
  - Pfizer Investigational Site, Cape Town
  - Pfizer Investigational Site, Gauteng
- South Korea (8):
  - Pfizer Investigational Site, Seo-gu, Busan
  - Pfizer Investigational Site, Jung-gu, Daegu
  - Pfizer Investigational Site, Anyang-si, Gyeonggi-do
  - Pfizer Investigational Site, Guri-si, Gyeonggi-do
  - Pfizer Investigational Site, Donggu, Kwangji
  - Pfizer Investigational Site, Gangnam-gu, Seoul
  - Pfizer Investigational Site, Yongdeungpo-gu, Seoul
  - Pfizer Investigational Site, Seoul
- Taiwan (4):
  - Pfizer Investigational Site, Niao-Sung Hsiang, Kaohsiung
  - Pfizer Investigational Site, Guei-Shan Shiang, Tau-Yuan Shian
  - Pfizer Investigational Site, Changhua
  - Pfizer Investigational Site, Taipei
- Thailand (3):
  - Pfizer Investigational Site, KHET Rajathevee, Bangkok
  - Pfizer Investigational Site, Bangkok
  - Pfizer Investigational Site, Chiang Mai
- Pfizer Investigational Site, Tunis, Tunisia
- Turkey (Türkiye) (9):
  - Pfizer Investigational Site, Cebeci, Ankara
  - Pfizer Investigational Site, Sihhiye, Ankara
  - Pfizer Investigational Site, Haydarpaşa, Istanbul
  - Pfizer Investigational Site, Alsancak, İzmir
  - Pfizer Investigational Site, Talas, Kayseri
  - Pfizer Investigational Site, Adana
  - Pfizer Investigational Site, Antalya
  - Pfizer Investigational Site, Diyarbakır
  - Pfizer Investigational Site, Istanbul
- United Arab Emirates (3):
  - Pfizer Investigational Site, Abu Dhabi
  - Pfizer Investigational Site, Dubai
  - Pfizer Investigational Site, Sharjah city
- Pfizer Investigational Site